CLINICAL TRIAL: NCT03574753
Title: A Phase II Study of ABBV-399 in Patients With C-Met Positive Stage IV or Recurrent Squamous Cell Lung Cancer (LUNG-MAP SUB-STUDY)
Brief Title: Lung-MAP S1400K: c-MET Positive
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S1400K
Record Dates: First submitted 2018-04-18; First posted 2018-07-02 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Squamous Cell Lung Carcinoma; Stage IV Squamous Cell Lung Carcinoma AJCC V7
MeSH Terms: interventions — telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABBV-399 (Experimental): C-MET overexpression is seen in 30% of patients with lung squamous cell carcinoma (SCCA). ABBV-399 (Process II) is a first-in-class antibody-drug conjugate (ADC) comprised of ABT-700, an anti-c-Met monoclonal antibody linked to monomethyl auristatin E (MMAE), which is a potent microtubule inhibitor. This delivers a direct anti-mitotic effect without relying on MET pathway inhibition.
  ABBV-399 will be administered intravenously on day 1 of each 21-day cycle. Treatment will continue in consenting patients until disease progression or intolerable toxicity.
  Interventions: Drug: ABBV-399

INTERVENTIONS:
Drug: ABBV-399 — ABBV-399 (Process II), 2.7 mg/kg IV over 30 ± 10 minutes, Day 1, Every 21 days

SUMMARY:
S1400K of Lung-MAP seeks to evaluate the overall response rate with ABBV-399 (Process II) in patients with c-MET positive SCCA.

S1400K is a biomarker-driven study for patients with Stage IV or recurrent squamous cell lung cancer, who have c-MET positive squamous cell tumors.

ELIGIBILITY:
•Patients must meet all SCREENING/PRE-SCREENING and SUB-STUDY REGISTRATION COMMON ELIGIBILITY CRITERIA as specified in S1400: A BIOMARKER-DRIVEN MASTER PROTOCOL FOR PREVIOUSLY TREATED SQUAMOUS CELL LUNG CANCER 5.1 Sub-Study Specific Disease Related Criteria

1. Patients must have been assigned to S1400I.
2. Patients must not have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell costimulation or immune checkpoint pathways.
3. Patients must not have an active, known, or suspected autoimmune disease. Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.

5.2 Sub-Study Specific Clinical/Laboratory Criteria

1. Patients must not have any known allergy or reaction to any component of the nivolumab and ipilimumab formulations.
2. Patients must not have received systemic treatment with corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days prior to sub-study registration. Inhaled or topical steroids, and adrenal replacement doses <= 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease.
3. Patients must not have a known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection. Patients with a positive hepatitis C antibody with a negative viral load are allowed. [This criterion replaces common eligibility criteria in Section 5.3m.]
4. Patients must not have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). [This criterion replaces common eligibility criteria in Section 5.3n.]
5. Patients must not have interstitial lung disease that is symptomatic or disease that may interfere with the detection or management of suspected drug-related pulmonary toxicity.
6. Patients must also be offered participation in banking for future use of specimens as described in Section 15.0.
7. Patients must have a Lipase, Amylase, TSH with reflex Free T3/T4 performed within 7 days prior to sub-study registration. Additional timepoints are noted in Section 9.0, Study Calendar. [Note: For the Canadian sites, testing for lipase only is acceptable.]
8. Patients must not have any Grade III/IV cardiac disease as defined by the New York Heart Association Criteria (i.e., patients with cardiac disease resulting in marked limitation of physical activity or resulting in inability to carry on any physical activity without discomfort), unstable angina pectoris, and myocardial infarction within 6 months, or serious uncontrolled cardiac arrhythmia (see Section 18.1b).

   1. Patients with a history of congestive heart failure (CHF) or at risk because of underlying cardiovascular disease or exposure to cardiotoxic drug should have an EKG and echocardiogram performed to evaluate cardiac function as clinically indicated.
   2. Patients with evidence of congestive heart failure (CHF), myocardial infarction (MI), cardiomyopathy, or myositis should have a cardiac evaluation including lab tests and cardiology consultations as clinically indicated including EKG, CPK, troponin, and echocardiogram.
9. Patients who can complete PRO forms in English are required to complete a pre-study S1400I Patient Reported Outcomes (PRO) Questionnaire and a pre-study S1400I EQ-5D Questionnaire within 14 days prior to registration (see Section 18.2 of S1400I). NOTE: Patients enrolled to S1400I prior to 9/1/2016 are not eligible for the PRO study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Waqar SN, Redman MW, Arnold SM, Hirsch FR, Mack PC, Schwartz LH, Gandara DR, Stinchcombe TE, Leighl NB, Ramalingam SS, Tanna SH, Raddin RS, Minichiello K, Bradley JD, Kelly K, Herbst RS, Papadimitrakopoulou VA. A Phase II Study of Telisotuzumab Vedotin in Patients With c-MET-positive Stage IV or Recurrent Squamous Cell Lung Cancer (LUNG-MAP Sub-study S1400K, NCT03574753). Clin Lung Cancer. 2021 May;22(3):170-177. doi: 10.1016/j.cllc.2020.09.013. Epub 2020 Oct 14. PMID 33221175

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants were enrolled, but 5 were ineligible. Thus 23 participants were eligible.
Groups:
- ABBV-399: C-MET overexpression is seen in 30% of participants with lung squamous cell carcinoma (SCCA). ABBV-399 (Process II) is a first-in-class antibody-drug conjugate (ADC) comprised of ABT-700, an anti-c-Met monoclonal antibody linked to monomethyl auristatin E (MMAE), which is a potent microtubule inhibitor. This delivers a direct anti-mitotic effect without relying on MET pathway inhibition.
  ABBV-399 will be administered intravenously on day 1 of each 21-day cycle. Treatment will continue in consenting patients until disease progression or intolerable toxicity.
  ABBV-399: ABBV-399 (Process II), 2.7 mg/kg IV over 30 ± 10 minutes, Day 1, Every 21 days
Period: Overall Study
Arm/Group | ABBV-399
Started | 23
Completed | 0
Not Completed | 23
Not completed — Adverse Event | 3
Not completed — Progression/relapse | 19
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABBV-399
Number analyzed (Participants) | 23
Age, Continuous [Median (Full Range); unit: years] | 65.3 [57.7 to 81.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21
  Asian | 2
  Hispanic | 0
Number of lines of prior therapy for stage IV SCC [Count of Participants; unit: Participants]
  0 | 7
  1 | 7
  2 | 5
  3 | 3
  4 | 1
ECOG performance status [Count of Participants; unit: Participants] — 0- fully active, able to carry out all pre-disease performance without restriction
  1- restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature
  Participants
    0 | 5
    1 | 18
Weight loss in the last 6 months [Count of Participants; unit: Participants]
  <5% | 17
  5%-<10% | 3
  10%-<20% | 3
Smoking status [Count of Participants; unit: Participants]
  Current | 7
  Former | 15
  Never | 1
Prior anti-programmed death-ligand (PD-L1) therapy [Count of Participants; unit: Participants]
  Yes | 12
  No | 11
Brain metastases at baseline [Count of Participants; unit: Participants]
  Yes | 2
  No | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate in Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA)
Description: The percentage of participants with confirmed and unconfirmed, partial response and complete response to treatment with ABBV-399 per Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1).
Time Frame: 11 months
Population: All eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-399
Number analyzed (Participants) | 23
percentage of participants | 9 [0 to 20]

2. Secondary Outcome: Investigator-assessed Progression-free Survival) in Immunotherapy-exposed and Relapsed Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA).
Description: Duration from date of sub-study registration to date of first documentation of progression, per RECIST 1.1, assessed by local review or symptomatic deterioration or death due to any cause.
Time Frame: up to 3 years post sub-study registration
Population: Eligible participants who had been on immunotherapy and relapsed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABBV-399
Number analyzed (Participants) | 12
months | 1.6 [1.4 to 3.0]

3. Secondary Outcome: Overall Survival (OS) in Immunotherapy-exposed and Relapsed Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA).
Description: Duration from date of sub-study registration (or date of screening/pre-screening registration if patient never enrolls in a sub-study) to date of death due to any cause
Time Frame: up to 3 years post sub-study registration
Population: Eligible participants who had been on immunotherapy and relapsed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABBV-399
Number analyzed (Participants) | 12
months | 4.8 [3.9 to 9.8]

4. Secondary Outcome: Overall Response Rate (ORR) in Immunotherapy-exposed and Relapsed Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA).
Description: as for outcome 1
Time Frame: Up to 3 years
Population: Eligible participants who had been on immunotherapy and relapsed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABBV-399
Number analyzed (Participants) | 12
percentage of participants | 0 [0 to 0]

5. Secondary Outcome: Investigator-assessed Progression-free Survival (IA-PFS) in Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA)
Description: as for outcome 2
Time Frame: Up to 3 years post sub-study registration
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABBV-399
Number analyzed (Participants) | 23
months | 2.4 [1.4 to 3.0]

6. Secondary Outcome: Overall Survival (OS) in Participants With c-Met Positive Lung Squamous Cell Carcinoma (SCCA)
Description: as for outcome 3
Time Frame: Up to 3 years post sub-study registration
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABBV-399
Number analyzed (Participants) | 23
months | 5.6 [3.9 to 9.5]

7. Secondary Outcome: Duration of Response (DoR)
Description: Duration from date of first documentation of response (complete or partial) to date of first documentation of progression assessed by local review or symptomatic deterioration, or death due to any cause among participants who achieve a complete or partial response.
Time Frame: Up to 3 years post sub-study registration
Population: Eligible participants who achieved complete or partial response.
Measure: Mean (Full Range); unit: months
Arm/Group | ABBV-399
Number analyzed (Participants) | 2
months | 8.9 [2.3 to 15.5]

8. Secondary Outcome: Number of Participants With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE Version 5.0 for serious adverse events only and CTCAE Version 4.0 for routine toxicity reporting. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post sub-registration
Population: Participants who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Groups:
- ABBV-399: C-MET overexpression is seen in 30% of participants with lung squamous cell carcinoma (SCCA). ABBV-399 (Process II) is a first-in-class antibody-drug conjugate (ADC) comprised of ABT-700, an anti-c-Met monoclonal antibody linked to monomethyl auristatin E (MMAE), which is a potent microtubule inhibitor. This delivers a direct anti-mitotic effect without relying on MET pathway inhibition.
  ABBV-399 will be administered intravenously on day 1 of each 21-day cycle. Treatment will continue in consenting patients until disease progression or intolerable toxicity.
  ABBV-399: ABBV-399 (Process II), 2.7 mg/kg IV over 30 ± 10 minutes, Day 1, Every 21 daysXXX
Arm/Group | ABBV-399
Number analyzed (Participants) | 23
Participants
  Anemia | 1
  Anorexia | 1
  Aspartate aminotransferase increased | 1
  Blood bilirubin increased | 1
  Bronchopulmonary hemorrhage | 1
  Cardiac arrest | 1
  Dehydration | 1
  Fatigue | 2
  Febrile neutropenia | 1
  Hypocalcemia | 1
  Hypokalemia | 1
  Hyponatremia | 1
  Hypophosphatemia | 2
  Lymphocyte count decreased | 1
  Nausea | 1
  Neutrophil count decreased | 1
  Peripheral sensory neuropathy | 1
  Pneumonitis | 2
  Respiratory failure | 1
  Urinary tract infection | 1
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post sub-study registration
Description: 23 eligible participants that received protocol therapy were assessed for AEs.
Arm/Group | ABBV-399
All-Cause Mortality (participants affected / at risk) | 17/23
Serious Adverse Events (participants affected / at risk) | 10/23
Other Adverse Events (participants affected / at risk) | 22/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABBV-399 (N=23)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Lung infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Nervous system disorders-Other (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABBV-399 (N=23)
Anemia (Blood and lymphatic system disorders) | 12
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Endocrine disorders-Other (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eye disorders-Other (Eye disorders) | 1
Watering eyes (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 9
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Esophageal pain (Gastrointestinal disorders) | 1
Esophageal stenosis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomach pain (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Chills (General disorders) | 4
Edema limbs (General disorders) | 3
Fatigue (General disorders) | 11
Flu like symptoms (General disorders) | 1
General disorders and admin site conditions - Other (General disorders) | 1
Non-cardiac chest pain (General disorders) | 4
Pain (General disorders) | 3
Infections and infestations-Other (Infections and infestations) | 2
Lung infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 3
Alanine aminotransferase increased (Investigations) | 3
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
GGT increased (Investigations) | 8
Investigations-Other (Investigations) | 4
Lymphocyte count decreased (Investigations) | 8
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 19
Hypocalcemia (Metabolism and nutrition disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 2
Dysphasia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Nervous system disorders-Other (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Renal and urinary disorders-Other (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03574753/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/53/NCT03574753/ICF_001.pdf